CLINICAL TRIAL: NCT03117049
Title: A Multicenter, Randomized, Double-Blind Trial in Subjects With Non-Squamous Non-Small Cell Lung Cancer (TASUKI-52)
Brief Title: Study of ONO-4538 in Non-Squamous Non-Small Cell Lung Cancer (TASUKI-52)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ONO-4538-52
Record Dates: First submitted 2017-04-12; First posted 2017-04-17 (Actual); Results first posted 2022-04-26 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Carboplatin; Paclitaxel; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ONO-4538 group (Experimental): ONO-4538: 360 mg solution intravenously for 30 min in every 3 weeks until RECIST 1.1 defined PD, unacceptable toxicity, or withdrawal of consent.
  Chemotherapy: Carboplatin at AUC 6 and Paclitaxel at 200 mg/m2 intravenously in every 3 weeks for up to 4 cycles and if deemed safe, Carboplatin and Paclitaxel may continue for up to a maximum of 6 cycles until RECIST 1.1 defined PD, unacceptable toxicity, or withdrawal of consent. Bevacizumab at 15 mg/kg intravenously in every 3 weeks until RECIST 1.1 defined PD, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: ONO-4538; Drug: Carboplatin; Drug: Paclitaxel; Drug: Bevacizumab
- Placebo group (Placebo Comparator): Placebo: Placebo solution intravenously for 30 min in every 3 weeks until RECIST 1.1 defined PD, unacceptable toxicity, or withdrawal of consent.
  Chemotherapy: Carboplatin at AUC 6 and Paclitaxel at 200 mg/m2 intravenously in every 3 weeks for up to 4 cycles and if deemed safe, Carboplatin and Paclitaxel may continue for up to a maximum of 6 cycles until RECIST 1.1 defined PD, unacceptable toxicity, or withdrawal of consent. Bevacizumab at 15 mg/kg intravenously in every 3 weeks until RECIST 1.1 defined PD, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Bevacizumab; Drug: Placebo

INTERVENTIONS:
Drug: ONO-4538 — 360 mg solution intravenously for 30 min in every 3 weeks until RECIST 1.1 defined PD, unacceptable toxicity, or withdrawal of consent.
  Arms: ONO-4538 group
Drug: Carboplatin — Carboplatin at AUC 6 and Paclitaxel at 200 mg/m2 intravenously in every 3 weeks for up to 4 cycles and if deemed safe, Carboplatin and Paclitaxel may continue for up to a maximum of 6 cycles until RECIST 1.1 defined PD, unacceptable toxicity, or withdrawal of consent.
Drug: Paclitaxel — Carboplatin at AUC 6 and Paclitaxel at 200 mg/m2 intravenously in every 3 weeks for up to 4 cycles and if deemed safe, Carboplatin and Paclitaxel may continue for up to a maximum of 6 cycles until RECIST 1.1 defined PD, unacceptable toxicity, or withdrawal of consent.
Drug: Bevacizumab — Bevacizumab at 15 mg/kg intravenously in every 3 weeks until RECIST 1.1 defined PD, unacceptable toxicity, or withdrawal of consent.
Drug: Placebo — Placebo solution intravenously for 30 min in every 3 weeks until RECIST 1.1 defined PD, unacceptable toxicity, or withdrawal of consent.
  Arms: Placebo group

SUMMARY:
The purpose of study is to compare the efficacy and safety of ONO-4538 in combination with carboplatin, paclitaxel, and bevacizumab (ONO-4538 group) to placebo in combination with carboplatin, paclitaxel, and bevacizumab (placebo group) in chemotherapy-naïve subjects with stage IIIB/IV or recurrent non-squamous non-small cell lung cancer unsuitable for radical radiation in a multicenter, randomized, double-blind study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically- or cytologically-confirmed non-squamous non-small cell lung cancer
* Subjects who received a diagnosis of stage IIIB/IV or recurrent non-squamous non-small cell lung cancer unsuitable for radical radiation according to the UICC-TNM Classification (7th edition) with no prior systemic anticancer therapy
* Subjects with at least one measurable lesion by radiographic tumor assessments per RECIST 1.1 criteria
* Subjects who are able to provide tumor tissue specimens.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 or 1

Exclusion Criteria:

* Subjects with known EGFR mutations, including deletions in exon 19 and exon 21 (L858R) substitution mutations.
* Subjects with known ALK translocations.
* Complication or history of severe hypersensitivity reactions to antibody products or platinum-containing compounds
* Subjects with autoimmune disease or known chronic or recurrent autoimmune disease.
* Subjects with multiple cancer.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2023-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Takahashi, Study Director — Ono Pharmaceutical Co. Ltd
Locations (135):
- Japan (110):
  - Aichi Clinical Site2, Nagoya, Aichi-ken
  - Aichi Clinical Site3, Nagoya, Aichi-ken
  - Aichi Clinical Site4, Nagoya, Aichi-ken
  - Aichi Clinical Site, Nagoya, Aichi-ken
  - Aichi Clinical Site, Toyoake, Aichi-ken
  - Aomori Clinical Site2, Hirosaki, Aomori
  - Aomori Clinical Site, Hirosaki, Aomori
  - Chiba Clinical Site, Yachiyo, Chiba
  - Ehime Clinical Site, Matsuyama, Ehime
  - Fukuoka Clinical Site, Iizuka, Fukuoka
  - Fukuoka Clinical Site, Kitakyushu, Fukuoka
  - Fukuoka Clinical Site, Koga, Fukuoka
  - Fukuoka Clinical Site, Kurume, Fukuoka
  - Fukushima Clinical Site, Kōriyama, Fukushima
  - Gunma Clinical Site, Ōta, Gunma
  - Gunma Clinical Site, Shibukawa, Gunma
  - Hokkaido Clinical Site, Asahikawa, Hokkaido
  - Hokkaido Clinical Site2, Sapporo, Hokkaido
  - Hokkaido Clinical Site, Sapporo, Hokkaido
  - Hyogo Clinical Site, Akashi, Hyōgo
  - Hyogo Clinical Site, Amagasaki, Hyōgo
  - Hyogo Clinical Site, Himeji, Hyōgo
  - Hyogo Clinical Site, Itami, Hyōgo
  - Hyogo Clinical Site, Kobe, Hyōgo
  - Hyogo Clinical Site, Nishinomiya, Hyōgo
  - Hyogo Clinical Site, Takarazuka, Hyōgo
  - Ibaraki Clinical Site, Higashiibaraki, Ibaraki
  - Ibaraki Clinical Site, Kasama, Ibaraki
  - Ibaraki Clinical Site, Tsuchiura, Ibaraki
  - Ishikawa Clinical Site2, Kanazawa, Ishikawa-ken
  - Ishikawa Clinical Site3, Kanazawa, Ishikawa-ken
  - Ishikawa Clinical Site, Kanazawa, Ishikawa-ken
  - Iwate Clinical Site, Morioka, Iwate
  - Kanagawa Clinical Site, Isehara, Kanagawa
  - Kanagawa Clinical Site2, Kawasaki, Kanagawa
  - Kanagawa Clinical Site, Kawasaki, Kanagawa
  - Kanagawa Clinical Site, Sagamihara, Kanagawa
  - Kanagawa Clinical Site2, Yokohama, Kanagawa
  - Kanagawa Clinical Site3, Yokohama, Kanagawa
  - Kanagawa Clinical Site, Yokohama, Kanagawa
  - Kumamoto Clinical Site, Kōshi, Kumamoto
  - Kyoto Clinical Site, Jōyō, Kyoto
  - Mie Clinical Site, Tsu, Mie-ken
  - Miyagi Clinical Site, Natori-shi, Miyagi
  - Miyagi Clinical Site, Sendai, Miyagi
  - Nagano Clinical Site, Matsumoto, Nagano
  - Nagasaki Clinical Site, Ōmura, Nagasaki
  - Nara Clinical Site, Ikoma, Nara
  - Niigata Clinical Site, Nagaoka, Niigata
  - Oita Clinical Site, Beppu, Oita Prefecture
  - Oita Clinical Site, Yufu, Oita Prefecture
  - Osaka Clinical Site, Habikino, Osaka
  - Osaka Clinical Site, Hirakata, Osaka
  - Osaka Clinical Site, Kishiwada, Osaka
  - Osaka Clinical Site, Sakai, Osaka
  - Osaka Clinical Site, Sayama, Osaka
  - Osaka Clinical Site, Toyonaka, Osaka
  - Osaka Clinical Site2, Osaka, Osaka Clinical Site
  - Saga Clinical Site, Ureshino, Saga-ken
  - Saitama Clinical Site, Hidaka, Saitama
  - Saitama Clinical Site, Kitaadachi-gun, Saitama
  - Shimane Clinical Site, Izumo, Shimane
  - Shizuoka Clinical Site, Hamamatsu, Shizuoka
  - Shizuoka Clinical Site, Sunto-gun, Shizuoka
  - Tokyo Clinical Site2, Bunkyo-ku, Tokyo
  - Tokyo Clinical Site, Bunkyo-ku, Tokyo
  - Tokyo Clinical Site2, Bunkyō-Ku, Tokyo
  - Tokyo Clinical Site2, Chuo-ku, Tokyo
  - Tokyo Clinical Site, Chuo-ku, Tokyo
  - Tokyo Clinical Site, Fuchū, Tokyo
  - Tokyo Clinical Site, Itabashi-ku, Tokyo
  - Tokyo Clinical Site, Kiyose, Tokyo
  - Tokyo Clinical Site, Koto-ku, Tokyo
  - Tokyo Clinical Site, Meguro City, Tokyo
  - Tokyo Clinical Site, Minato-ku, Tokyo
  - Tokyo Clinical Site, Mitaka-shi, Tokyo
  - Tokyo Clinical Site, Shibuya City, Tokyo
  - Tokyo Clinical Site2, Shinjuku-Ku, Tokyo
  - Tokyo Clinical Site3, Shinjuku-Ku, Tokyo
  - Tokyo Clinical Site, Shinjuku-ku, Tokyo
  - Tokyo Clinical Site, Tachikawa, Tokyo
  - Tottori Clinical Site, Yonago, Tottori
  - Yamaguchi Clinical Site, Iwakuni, Yamaguchi
  - Chiba Clinical Site2, Chiba
  - Chiba Clinical Site, Chiba
  - Fukui Clinical Site, Fukui
  - Fukuoka Clinical Site2, Fukuoka
  - Fukuoka Clinical Site3, Fukuoka
  - Fukuoka Clinical Site4, Fukuoka
  - Fukuoka Clinical Site, Fukuoka
  - Gifu Clinical Site2, Gifu
  - Gifu Clinical Site, Gifu
  - Hiroshima Clinical Site2, Hiroshima
  - Hiroshima Clinical Site, Hiroshima
  - Kochi Clinical Site, Kochi
  - Kumamoto Clinical Site, Kumamoto
  - Kyoto Clinical Site, Kyoto
  - Nagasaki Clinical Site, Nagasaki
  - Niigata Clinical Site2, Niigata
  - Niigata Clinical Site, Niigata
  - Okayama Clinical Site2, Okayama
  - Okayama Clinical Site, Okayama
  - Osaka Clinical Site3, Osaka
  - Osaka Clinical Site, Osaka
  - Oita Clinical Site, Ōita
  - Tokushima Clinical Site, Tokushima
  - Toyama Clinical Site2, Toyama
  - Toyama Clinical Site, Toyama
  - Wakayama Clinical Site, Wakayama
  - Yamaguchi Clinical Site, Yamaguchi
- South Korea (15):
  - Gangwon-Do Clinical Site, Wŏnju, Gangwon-do
  - Gyeonggi-do Clinical Site2, Seongnam-si, Gyeonggi-do
  - Gyeonggi-do Clinical Site, Seongnam-si, Gyeonggi-do
  - Gyeonggi-do Clinical Site, Suwon, Gyeonggi-do
  - Gyeongsangnam-do Clinical Site, Jinju, Gyeongsangnam-do
  - Chungcheongbuk-do Clinical Site, Cheongju-si, North Chungcheong
  - Busan Clinical Site, Busan
  - Daegu Clinical Site, Daegu
  - Incheon Clinical Site, Incheon
  - Seoul Clinical Site2, Seoul
  - Seoul Clinical Site3, Seoul
  - Seoul Clinical Site4, Seoul
  - Seoul Clinical Site5, Seoul
  - Seoul Clinical Site6, Seoul
  - Seoul Clinical Site, Seoul
- Taiwan (10):
  - Changhua Clinical Site, Changhua
  - Chiayi Clinical Site, Chiayi City
  - Kaohsiung Clinical Site2, Kaohsiung City
  - Kaohsiung Clinical Site3, Kaohsiung City
  - Kaohsiung Clinical Site, Kaohsiung City
  - Taichung Clinical Site, Taichung
  - Tainan Clinical Site, Tainan
  - Taipei Clinical Site2, Taipei
  - Taipei Clinical Site, Taipei
  - Taoyuan Clinical Site, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sugawara S, Lee JS, Kang JH, Kim HR, Inui N, Hida T, Lee KH, Yoshida T, Tanaka H, Yang CT, Inoue T, Nishio M, Goto Y, Tamura T, Yamamoto N, Yu CJ, Akamatsu H, Takahashi S, Nakagawa K. Plain language summary of TASUKI-52: A study looking at nivolumab plus platinum chemotherapy and bevacizumab as a combined treatment for people with advanced or recurrent nonsquamous non-small cell lung cancer (NSCLC). Future Oncol. 2026 Feb 4:1-13. doi: 10.1080/14796694.2026.2617855. Online ahead of print. PMID 41640231
- [Derived] Lee JS, Sugawara S, Kang JH, Kim HR, Inui N, Hida T, Lee KH, Yoshida T, Tanaka H, Yang CT, Inoue T, Nishio M, Goto Y, Tamura T, Yamamoto N, Yu CJ, Akamatsu H, Takahashi S, Nakagawa K. Four-Year Outcomes for Nivolumab With Chemotherapy and Bevacizumab in Patients With Nonsquamous NSCLC in the TASUKI-52. Cancer Sci. 2026 Jan 29. doi: 10.1111/cas.70330. Online ahead of print. PMID 41611341
- [Derived] Kim HR, Sugawara S, Lee JS, Kang JH, Inui N, Hida T, Lee KH, Yoshida T, Tanaka H, Yang CT, Nishio M, Ohe Y, Tamura T, Yamamoto N, Yu CJ, Akamatsu H, Takahashi S, Nakagawa K. First-line nivolumab, paclitaxel, carboplatin, and bevacizumab for advanced non-squamous non-small cell lung cancer: Updated survival analysis of the ONO-4538-52/TASUKI-52 randomized controlled trial. Cancer Med. 2023 Aug;12(16):17061-17067. doi: 10.1002/cam4.6348. Epub 2023 Aug 28. PMID 37641544

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ONO-4538 Group | Placebo Group
Started (Randomized) | 275 | 275
Completed (Continued at least one study treatment at the time of cut-off) | 74 | 44
Not Completed | 201 | 231
Not completed — Continued the follow-up period | 109 | 129
Not completed — Died | 82 | 93
Not completed — Consent withdrawal | 7 | 6
Not completed — Missing contact | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ONO-4538 Group | Placebo Group | Total
Number analyzed (Participants) | 275 | 275 | 550
Age, Continuous [Median (Full Range); unit: years] | 66 [27 to 85] | 66 [33 to 83] | 66 [27 to 85]
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 131 | 111 | 242
  65-74 years | 117 | 131 | 248
  >=75 years | 27 | 33 | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 69 | 139
  Male | 205 | 206 | 411
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 275 | 275 | 550
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Country [Count of Participants; unit: Participants]
  Japan | 188 | 183 | 371
  Korea | 62 | 63 | 125
  Taiwan | 25 | 29 | 54
ECOG Performance Score [Count of Participants; unit: Participants] — Interactive Web Response System source. Score 0 : Fully active, able to carry on all pre-disease performance without restriction, Score 1 : Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, eg, light house work, office work
  Participants
    0 | 129 | 128 | 257
    1 | 146 | 147 | 293
Smoking status [Count of Participants; unit: Participants] — Former smokers included anyone who had smoked even a small quantity of any tobacco and had stopped smoking at the time of screening. Current smokers are anyone who had a smoking habit of any tobacco regardless of smoking duration/quantity at the screening.
  Participants
    Never | 61 | 54 | 115
    Current | 18 | 21 | 39
    Former | 196 | 200 | 396
Staging (the UICC-TNM classification, 7th edition) [Count of Participants; unit: Participants] — Stage IIIB:T4(Tumor of any size that invades the mediastinum, heart, great vessels, trachea, recurrent laryngeal nerve, esophagus, vertebral body, carina, or with separate tumor nodules in a different ipsilateral lobe) and N2(Metastasis in ipsilateral mediastinal and/or subcarinal lymph node(s)), or N3(Metastasis in contralateral mediastinal, contralateral hilar, ipsilateral or contralateral scalene, or supraclavicular lymph node(s)) with any T Stage IV:Distant metastasis
  Participants
    Stage IIIB | 15 | 14 | 29
    Stage IV | 239 | 238 | 477
    Recurrent | 21 | 23 | 44
Metastasis [Count of Participants; unit: Participants]
  Bone | 56 | 83 | 139
  Liver | 19 | 20 | 39
  Brain | 36 | 41 | 77
PD-L1 expression levels [Count of Participants; unit: Participants] — Interactive Web Response System source. There were five patients with indeterminate PD-L1 expression levels in both arms.
  Participants
    <1% or indeterminate | 120 | 120 | 240
    1%-49% | 82 | 81 | 163
    >=50 | 73 | 74 | 147

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) as Assessed by the Independent Radiology Review Committee (IRRC)
Description: PFS (as assessed by the IRRC) will be calculated using the following formula : PFS (days) = "date when overall response is assessed as progressive disease (PD) or date of death (for any reason), whichever comes first" - "date of randomization" + 1. Please refer to the protocol, in this study, tumor response will be evaluated by CT, etc. according to the RECIST 1.1 criteria.
Time Frame: Approximately 32 months
Measure: Median (96.37% Confidence Interval); unit: months
Arm/Group | ONO-4538 Group | Placebo Group
Number analyzed (Participants) | 275 | 275
months | 12.1 [9.8 to 14.0] | 8.1 [7.0 to 8.5]
Statistical Analysis 1: Comparison: ONO-4538 Group vs Placebo Group; Test type: Superiority; p < 0.0001, Stratified log-rank test; Hazard Ratio (HR) = 0.56, 96.37% CI 2-sided [0.43 to 0.71]

2. Secondary Outcome: Overall Survival (OS)
Time Frame: Approximately 32 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ONO-4538 Group | Placebo Group
Number analyzed (Participants) | 275 | 275
months | 25.4 [21.8 to NA] — The Upper Limit has not been reached due to insufficient number of participants with events. | 24.7 [20.2 to NA] — The Upper Limit has not been reached due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: ONO-4538 Group vs Placebo Group; Test type: Superiority; Stratified hazard ratio = 0.85, 95% CI 2-sided [0.63 to 1.14]

3. Secondary Outcome: Objective Response Rate (ORR [as Assessed by the IRRC])
Description: ORR represents the proportion of subjects whose best overall response was assessed as complete response (CR) or partial response (PR). Please refer to the protocol, in this study, tumor response will be evaluated by CT, etc. according to the RECIST 1.1 criteria.
Time Frame: Approximately 32 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ONO-4538 Group | Placebo Group
Number analyzed (Participants) | 275 | 275
percentage of participants | 61.5 [55.4 to 67.2] | 50.5 [44.5 to 56.6]
Statistical Analysis 1: Comparison: ONO-4538 Group vs Placebo Group; Test type: Superiority; Odds Ratio (OR) = 1.55, 95% CI 2-sided [1.11 to 2.17]

4. Secondary Outcome: Disease Control Rate (DCR [as Assessed by the IRRC])
Description: DCR represents the proportion of subjects whose best overall response was assessed as CR, PR, or stable disease (SD). Please refer to the protocol, in this study, tumor response will be evaluated by CT, etc. according to the RECIST 1.1 criteria.
Time Frame: Approximately 32 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ONO-4538 Group | Placebo Group
Number analyzed (Participants) | 275 | 275
percentage of participants | 87.3 [82.7 to 91.0] | 89.8 [85.6 to 93.1]
Statistical Analysis 1: Comparison: ONO-4538 Group vs Placebo Group; Test type: Superiority; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.46 to 1.31]

5. Secondary Outcome: Duration of Response (DOR [as Assessed by the IRRC])
Description: The lower and upper limits of 95% CI for the median are censored value in the both groups.
Time Frame: Approximately 32 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ONO-4538 Group | Placebo Group
Number analyzed (Participants) | 275 | 275
months | 11.0 [1.1 to 25.8] | 7.0 [1.2 to 26.0]

6. Secondary Outcome: Best Overall Response (BOR [as Assessed by the IRRC])
Time Frame: Approximately 32 months
Population: For best overall response to be assessed as stable disease in this study, at least one stable disease or better rather than progressive disease on or after day 43 should be obtained.
Measure: Count of Participants; unit: Participants
Arm/Group | ONO-4538 Group | Placebo Group
Number analyzed (Participants) | 275 | 275
Participants
  Complete response | 14 | 8
  Partial response | 155 | 131
  Stable disease | 71 | 108
  Progressive disease | 5 | 11
  Not evaluable | 30 | 17

ADVERSE EVENTS:
Time Frame: For each randomised subject, adverse events(AEs) were collected from the start date of administration of the investigational product to 30 days after the last dose of any of the study treatment (The maximum was about 30 months). Drug-related AEs or AEs leading to discontinuation reported at the start of follow-up should be investigated at appropriate intervals until no further follow-up is required because the events have resolved or are resolving, or the symptoms become stable.
Description: All-Cause Mortality indicates the number of patients who died by any cause (e.g. Primary disease) from the start of the study to data cut off (approximately 32 months).
  Overall Number of Participants Analyzed in efficacy and All-cause Mortality is among ITT, whereas the risk population (AEs) is among SAF. Above is the reason of the gap b/w 275 and 273.
  ITT: consist of all randomized subjects. SAF: consist of all subjects who received the investigational product or chemotherapy at least once.
Arm/Group | ONO-4538 Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 82/275 | 93/275
Serious Adverse Events (participants affected / at risk) | 154/273 | 118/275
Other Adverse Events (participants affected / at risk) | 271/273 | 274/275
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ONO-4538 Group (N=273) | Placebo Group (N=275)
Anaemia (Blood and lymphatic system disorders) | 5 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 27 | 12
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Splenic haemorrhage (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 2
Angina unstable (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 7 | 1
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 1 | 0
Hypopituitarism (Endocrine disorders) | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0
Anal ulcer (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 8 | 1
Colitis microscopic (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 1
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 3
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Pancreatic fistula (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 1 | 0
Rectal prolapse (Gastrointestinal disorders) | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 2 | 3
Chest pain (General disorders) | 0 | 1
Death (General disorders) | 1 | 1
Fatigue (General disorders) | 0 | 1
Haemorrhagic cyst (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Pyrexia (General disorders) | 16 | 4
Sudden death (General disorders) | 2 | 1
Biloma (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 2 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 4 | 1
Anaphylactic reaction (Immune system disorders) | 2 | 1
Anal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 3 | 0
Bronchitis (Infections and infestations) | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 2 | 0
Enteritis infectious (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis bacterial (Infections and infestations) | 1 | 0
Haematoma infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 2
Infectious pleural effusion (Infections and infestations) | 1 | 0
Large intestine infection (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 1 | 1
Osteomyelitis acute (Infections and infestations) | 1 | 0
Otitis media chronic (Infections and infestations) | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 0 | 1
Pleural infection bacterial (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 21 | 15
Pneumonia bacterial (Infections and infestations) | 2 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 0 | 1
Pseudomonal bacteraemia (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 2 | 3
Septic shock (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Post procedural fistula (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
Angiocardiogram (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 6 | 0
Platelet count decreased (Investigations) | 0 | 1
Weight increased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 5 | 8
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Fulminant type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small intestine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1
Brain stem infarction (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 2 | 2
Depressed level of consciousness (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 1
Epilepsy (Nervous system disorders) | 1 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2
Polyneuropathy (Nervous system disorders) | 1 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 0
Postresuscitation encephalopathy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 2 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 5 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 9 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 4 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 3 | 2
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ONO-4538 Group (N=273) | Placebo Group (N=275)
Anaemia (Blood and lymphatic system disorders) | 88 | 102
Febrile neutropenia (Blood and lymphatic system disorders) | 19 | 15
Leukopenia (Blood and lymphatic system disorders) | 26 | 19
Neutropenia (Blood and lymphatic system disorders) | 52 | 38
Thrombocytopenia (Blood and lymphatic system disorders) | 17 | 21
Tinnitus (Ear and labyrinth disorders) | 1 | 7
Adrenal insufficiency (Endocrine disorders) | 9 | 5
Hyperthyroidism (Endocrine disorders) | 15 | 4
Hypothyroidism (Endocrine disorders) | 27 | 8
Cataract (Eye disorders) | 2 | 6
Abdominal distension (Gastrointestinal disorders) | 7 | 4
Abdominal pain (Gastrointestinal disorders) | 9 | 11
Abdominal pain upper (Gastrointestinal disorders) | 13 | 8
Cheilitis (Gastrointestinal disorders) | 6 | 2
Constipation (Gastrointestinal disorders) | 150 | 134
Dental caries (Gastrointestinal disorders) | 12 | 2
Diarrhoea (Gastrointestinal disorders) | 81 | 66
Dry mouth (Gastrointestinal disorders) | 7 | 1
Dyspepsia (Gastrointestinal disorders) | 14 | 13
Gastritis (Gastrointestinal disorders) | 8 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 8
Gingival pain (Gastrointestinal disorders) | 8 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 5 | 6
Haemorrhoids (Gastrointestinal disorders) | 7 | 10
Nausea (Gastrointestinal disorders) | 86 | 100
Periodontal disease (Gastrointestinal disorders) | 5 | 8
Stomatitis (Gastrointestinal disorders) | 60 | 59
Vomiting (Gastrointestinal disorders) | 32 | 28
Asthenia (General disorders) | 8 | 13
Fatigue (General disorders) | 24 | 31
Infusion site extravasation (General disorders) | 9 | 7
Malaise (General disorders) | 72 | 78
Oedema peripheral (General disorders) | 16 | 13
Pain (General disorders) | 7 | 5
Pyrexia (General disorders) | 64 | 41
Hepatic function abnormal (Hepatobiliary disorders) | 20 | 9
Bronchitis (Infections and infestations) | 9 | 8
Conjunctivitis (Infections and infestations) | 5 | 6
Gingivitis (Infections and infestations) | 5 | 9
Herpes zoster (Infections and infestations) | 5 | 7
Influenza (Infections and infestations) | 7 | 4
Nasopharyngitis (Infections and infestations) | 22 | 19
Paronychia (Infections and infestations) | 3 | 7
Periodontitis (Infections and infestations) | 12 | 7
Pharyngitis (Infections and infestations) | 13 | 9
Pneumonia (Infections and infestations) | 17 | 13
Rhinitis (Infections and infestations) | 6 | 6
Upper respiratory tract infection (Infections and infestations) | 24 | 18
Urinary tract infection (Infections and infestations) | 4 | 10
Infusion related reaction (Injury, poisoning and procedural complications) | 9 | 6
Alanine aminotransferase increased (Investigations) | 33 | 35
Amylase increased (Investigations) | 10 | 0
Aspartate aminotransferase increased (Investigations) | 37 | 28
Blood alkaline phosphatase increased (Investigations) | 10 | 12
Blood bilirubin increased (Investigations) | 7 | 8
Blood creatine phosphokinase increased (Investigations) | 4 | 10
Blood creatinine increased (Investigations) | 22 | 18
Gamma-glutamyltransferase increased (Investigations) | 23 | 11
Lymphocyte count decreased (Investigations) | 15 | 9
Neutrophil count decreased (Investigations) | 117 | 141
Platelet count decreased (Investigations) | 62 | 67
Weight decreased (Investigations) | 23 | 16
White blood cell count decreased (Investigations) | 94 | 99
Decreased appetite (Metabolism and nutrition disorders) | 98 | 108
Dehydration (Metabolism and nutrition disorders) | 4 | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 12 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 13 | 14
Hyperuricaemia (Metabolism and nutrition disorders) | 11 | 11
Hypoalbuminaemia (Metabolism and nutrition disorders) | 18 | 15
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 11
Hyponatraemia (Metabolism and nutrition disorders) | 14 | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 72 | 84
Arthritis (Musculoskeletal and connective tissue disorders) | 5 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 26 | 19
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 6
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 76 | 92
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 16
Dizziness (Nervous system disorders) | 10 | 21
Dysgeusia (Nervous system disorders) | 33 | 20
Headache (Nervous system disorders) | 35 | 28
Hypoaesthesia (Nervous system disorders) | 10 | 12
Neuropathy peripheral (Nervous system disorders) | 59 | 64
Paraesthesia (Nervous system disorders) | 15 | 18
Peripheral sensory neuropathy (Nervous system disorders) | 121 | 116
Somnolence (Nervous system disorders) | 1 | 7
Delirium (Psychiatric disorders) | 4 | 7
Insomnia (Psychiatric disorders) | 45 | 49
Dysuria (Renal and urinary disorders) | 2 | 6
Proteinuria (Renal and urinary disorders) | 67 | 74
Renal impairment (Renal and urinary disorders) | 6 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 34
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 8 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 51 | 48
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 11 | 12
Hiccups (Respiratory, thoracic and mediastinal disorders) | 45 | 36
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 | 13
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 13 | 11
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 16
Alopecia (Skin and subcutaneous tissue disorders) | 143 | 150
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 23 | 17
Drug eruption (Skin and subcutaneous tissue disorders) | 7 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 32 | 24
Erythema (Skin and subcutaneous tissue disorders) | 6 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 61 | 48
Rash (Skin and subcutaneous tissue disorders) | 96 | 48
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 29 | 14
Urticaria (Skin and subcutaneous tissue disorders) | 16 | 7
Hypertension (Vascular disorders) | 74 | 89
Hypotension (Vascular disorders) | 7 | 9
Vasculitis (Vascular disorders) | 7 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this tiral prior to submission for publication/presentation.

DOCUMENTS (2):
  • Study Protocol (2019-10-17): https://cdn.clinicaltrials.gov/large-docs/49/NCT03117049/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/49/NCT03117049/SAP_001.pdf